CLINICAL TRIAL: NCT01420133
Title: Is a Low Salt Diet and Low Sugar Content Necessary When Corticosteroid Treatment is Prescribed?
Brief Title: Is a Diet Necessary When Corticosteroid Treatment is Prescribed?
Acronym: Cortisel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: K080906; AFSSAPS (Other: 2010-A01439-30)
Record Dates: First submitted 2011-06-23; First posted 2011-08-19 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Autoimmune Diseases; Asthma
Keywords: Corticosteroids; Diet low in sugar and salt; Dermatological disease; Corticosteroids Allergy; 3 Months
MeSH Terms: conditions — Autoimmune Diseases; Asthma; Skin Diseases | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal regimen (Experimental): without special regimen for corticosteroid therapy
  Interventions: Other: Regimen
- Standard arm (Active Comparator): with diet low in salt and sugar
  Interventions: Other: Standard regimen

INTERVENTIONS:
Other: Regimen — regimen normal in salt and sugar
  Arms: Normal regimen
Other: Standard regimen — with diet low in salt and sugar
  Arms: Standard arm

SUMMARY:
Few recommendations concerning the diet and dosage to be administered to patients treated with corticosteroids are established.

It therefore seems important to study prospectively the indication of a diet low in salt and sugar in patients undergoing corticosteroid therapy, to record side effects observed and to measure their frequency.

DETAILED DESCRIPTION:
In the French clinical patterns governing the prescription of corticosteroids, it is customary to prescribe a diet low in salt and low in sugar. This dietary prescription is based on the interest of any diet to prevent the occurrence of side effects of steroids such as hypertension, obesity, diabetes and congestive heart.

However, there is no specific dietary requirements in other European countries. This lack of recommendations is based on the fact that there is no evidence that a strict diet reduces the side effects of steroids on the one hand and secondly, that the quality of life of patients undergoing a diet low in salt and low in sugars affects their quality of life. In addition, no prospective study has helped to establish the frequency of side effects of corticosteroids depending on dose and duration of treatment.

The investigators therefore propose to study whether a diet intervention with low salt or low sugar during a prolonged corticosteroid treatment has any interest and effectively reduces the frequency and severity of side effects.

The investigators propose that all parameters being equal, to randomize the diet of patients started on steroids for a predictable period of 3 months minimum for a dose greater than 20 mg per day. One group will observe the low-salt diet, low in sugar and the other will follow a normal diet. The assessment will be made after 1 year, even if steroid treatment is continued beyond.

ELIGIBILITY:
Inclusion criteria :

* Age > 18 years
* All patients for whom corticoids initially prescribed at a dose > 20 mg per 24 hours, during a period of 3 months minimum
* Corticotherapy should be prescribed per os and continuously. (Alternating doses of corticoids, sequential intramuscular or intravenous injection of corticoids are not allowed in this clinical trial)
* All diseases requiring corticotherapy may be subject to this clinical trial. The main pathologies will be systemic autoimmune diseases, asthma or chronic skin diseases justifying prolonged oral corticotherapy.
* Time between first corticoids delivery and randomization < 1 month
* Patient who gave his non-opposition

Note: Depending on their health condition, patient may receive one or more intravenous injections of methylprednisolone (until 3 injections), before the beginning of oral corticotherapy.

Exclusion criteria :

* Age < 18 years or whose disability warrants a guardianship
* All patients for whom corticoids prescribed <20 mg per 24 hours or for an expected period <3 months
* Intramuscular or intravenous sequential corticoids delivery, without associated per os corticoids.
* Any corticotherapies other than prednisone, prednisolone or methylprednisolone.
* Any corticotherapies with alternating doses
* Intravenous or intramuscular injection corticotherapy
* Patient who received corticoids at a dose >20 mg / day, during 3 last years
* Allergy, hypersensitivity or cons-indication to corticoids
* The existence of diabetes before corticotherapy, because pre-existing diabetes requires specific follow-up treatment, such as sugars restrictions
* Uncontrolled hypertension (SBP ≥ 180mHg or DBP ≥ 110mHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cumulative number of clinical events recorded during the study, per randomization group | 24 months
  Cumulative number of the following clinical events recorded during the study, per randomization group:
  * Weight gain between study entry and the end of it
  * Significant rise in blood pressure between study entry and the end of it
  * Development of diabetes requiring treatment, whether prescribed oral or injectable and defined by international criteria of fasting glucose> 7 mmol / fasting twice or post prandial > 11,1 mmol/l twice
  * Occurrence of heart failure
Observance of the diet low in salt and sugar will be estimated by patient questionnaire and diary | 12 months
Tolerance of the diet low in salt and sugar will be estimated by patient questionnaire and diary | 12 months
Observance of the diet low in salt and sugar will be estimated by patient questionnaire and diary | 6 months
Tolerance of the diet low in salt and sugar will be estimated by patient questionnaire and diary | 6 months

SECONDARY OUTCOMES:
Sides effects of corticosteroids therapy | 24 months
  frequency of sides effects
Impaired glucide metabolism | 24 months
  surveillance of creatininemia, urinary and serum electrolytes changes
  * Glucose regulation change observed by blood glucose, insulin, QUICKI and OGTT tests performed at the beginning and the end of the study.
  * Evaluation of the pancreatic beta cell function (HOMA-B%) estimated as Matthews et al., 1985 done.

CONTACTS AND LOCATIONS:
Overall Officials: Loic Guillevin, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Jessie Aouizerate, MD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Cochin Hospital, Paris, France